CLINICAL TRIAL: NCT07297186
Title: A Randomized, Blinded, Parallel Positive-controlled Clinical Trial of Sabin Strain Inactivated Poliovirus Vaccine (Vero Cell) Conducted in Healthy Infants Aged Two Months.
Brief Title: Phase III Clinical Trial of Sabin Strain Inactivated Poliovirus Vaccine (Vero Cell)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017L00935
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 600 participants
  Interventions: Biological: sIPV
- control group (Active Comparator): 600 participants
  Interventions: Biological: wIPV

INTERVENTIONS:
Biological: sIPV — sIPVs were developed by Biominhai (Beijing Minhai Biotechnology Co. Ltd.)
  Arms: study group
Biological: wIPV — wIPVs were developed by Sanofi Pasteur
  Arms: control group

SUMMARY:
The study aimed to evaluate the safety and immunogenicity of a Sabin strain-based inactivated polio vaccine in infants aged two months (60~89 days).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy permanent residents aged 2 months (60~89 days);
2. Infant's legal guardians agree to sign the informed consent forms voluntarily;
3. Infant's legal guardians are able to comply with the requirements of the clinical trial protocol;
4. Armpit temperature ≤ 37.0 ℃

Exclusion Criteria:

1. preterm birth (gestational age < 37 weeks);
2. the presence of congenital malformations, developmental disorders, genetic defects, or severe malnutrition;
3. had a history of poliomyelitis;
4. had a personal or family history of allergy, convulsions, epilepsy, encephalopathy, or psychiatric disorders;
5. had known hypersensitivity to any component of the study vaccine or a history of severe allergic reaction (e.g., anaphylaxis) to any previous vaccination;
6. had immunodeficiency or receipt of immunosuppressive therapy;
7. diagnosed coagulation disorders (including factor deficiencies, coagulopathies, platelet abnormalities) or evidence of significant bruising/bleeding diathesis;
8. had known or investigator-suspected concurrent acute or active chronic diseases (including respiratory, cardiovascular, hepatic, renal, or dermatological conditions) or acute infection, or maternal HIV infection;
9. occurrence of fever (axillary temperature ≥ 38.0 °C) within the 3 days preceding enrollment;
10. had acute illness requiring systemic antibiotic or antiviral treatment within the 7 days preceding enrollment;
11. administration of blood products within the 3 months preceding enrollment;
12. had receipt of any live attenuated vaccine within the 14 days preceding enrollment;
13. had receipt of any inactivated or subunit vaccine within the 7 days preceding enrollment;
14. had recent administration of any other experimental product and any other condition deemed by the investigator as potentially interfering with the assessment of trial outcomes.

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
the seroconversion rates of poliovirus type I, type II and type III neutralizing antibodies | 30 days after the primary immunization

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No